CLINICAL TRIAL: NCT06726434
Title: Evaluation of Percutaneous Cryoneurotomy Compared to Surgical Open Neurotomy for the Management of Equinovarus Foot Deformity in Patients With Refractory Lower Limb Spasticity After Stroke: a Multicenter, Randomized Controlled, Non-inferiority Trial
Brief Title: Evaluation of Percutaneous Cryoneurotomy Compared to Surgical Open Neurotomy for the Management of Equinovarus Foot Deformity in Patients With Refractory Lower Limb Spasticity After Stroke
Acronym: CRYOSTROKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRYOSTROKE
Record Dates: First submitted 2024-11-22; First posted 2024-12-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Equinovarus Foot; Refractory Lower Limb Spasticity
Keywords: surgical neurotomy; CryoNeurotomy; spasticity; cryoneurolysis; percutaneous cryoneurolysis
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CryoNeurotomy (CN) (Experimental): Cryoneurotomy procedure
  Interventions: Procedure: Cryoneurotomy (CN)
- Surgical neurotomy (SN) (Active Comparator): Surgical neurotomy procedure
  Interventions: Procedure: Surgical neurotomy (SN)

INTERVENTIONS:
Procedure: Surgical neurotomy (SN) — Surgical neurotomy will be performed under general anesthesia according to the previous description. Muscle relaxant drugs will not be used in order to prevent any interference with the intraoperative electrical stimulation.
  The patient will be placed in a prone position and a vertical cutaneous incision will be made at the popliteal fossa location.
  The tibial nerve will be dissected and the motor nerve branches of the soleus, gastrocnemius, tibialis posterior and flexor hallucis longus will be identified with intraoperative tripolar electrical stimulation. The selected motor nerve branches will be partially sectioned over a 5mm length under the microscope. The extent of nerve section will be determined according to the degree of spasticity and to the intraoperative residual muscular contraction under electrical stimulation
  Arms: Surgical neurotomy (SN)
Procedure: Cryoneurotomy (CN) — After the use of an aseptic technique with 2% chlorhexidine, betadine application and a local anesthesia with lidocaine 1% (3ml), percutaneous cryoneurotomy will be performed with METRUM CRYOFLEX device guided by ultrasound with 1.2mm cryoprobe at -89°C placed through a #16 angio guide. Electrical stimulation will be performed to confirm tibial nerve contact at 0.8 mV.
  The ice ball will be repositioned to two spots along the nerve. Each lesion will be treated for 2min cryoneurolysis at -89°C, followed by 2min without freezing (passive defreezing period) and 2min of cryoneurolysis at -89°C, based on cryotherapy for pain management.
  Arms: CryoNeurotomy (CN)

SUMMARY:
CRYOSTROKE study is designed :

* to compare the efficacy and safety of percutaneous CryoNeurotomie (CN) versus surgical neurotomy (SN) on spasticity, 90 days after intervention, in post-stroke patients presenting with spastic equinovarus foot and,
* to ensure that potential clinical effect/safety remain stable within time, with a 12-month follow-up.

DETAILED DESCRIPTION:
Stroke, arising from cerebral vascular hemorrhage or ischemia, represents a major health-care problem affecting more than 140,000 persons in France every year. One of the major concerns after stroke is impairment of the pyramidal tract and parapyramidal fibers, resulting in upper motor neuron syndrome and spasticity. Up to 20% to 40% of stroke survivors develop spasticity, which dramatically impacts health status, pain, functional capacity, and ultimately, quality of life. Spastic equinovarus foot (SEF) is the most common deformity due to lower limb spasticity and is defined as a combination of an abnormal plantar-flexion, inversion and adduction of the foot. Consequently, SEF severely impairs walking capability and mobility, impacting daily life activities and restricting social participation. In addition to therapeutical physical rehabilitation programs, two main treatments can be proposed. First, SEF can be initially treated with focal botulinum toxin injections that for reducing spasticity. However, botulinum toxin injections are effective for only a limited period of time, and iterative reinjections are required. Second, permanent treatment of spasticity can be achieved by surgical neurotomy. This procedure, variably combined with muscle and tendon lengthening in the event of associated retractions, can be considered as the long-term radical and effective gold standard, but at the price of surgical invasiveness and complications.

A recent alternative allowing for both permanent treatment and a minimally invasive approach has been introduced: "percutaneous cryoneurotomy". While this approach has provided promising results, as shown in multiple case reports, its efficacy has yet to be determined in a randomized control study.

CryoNeurotomy (CN) was first performed and developed in daily practice for the upper limb. Through a mentoring process, a feasibility study was performed on cadavers and transposed the technique to human procedures in a pilot study. The results from the first patients, with a 90-day follow-up period, are promising, with decreased spasticity and significantly increased walking capabilities. Major potential advantages of percutaneous CN compared to surgical neurotomy were identified, such as minimal skin incision, faster procedure, far less invasiveness of muscle tissue and adjacent neuro-vascular structures, particularly a decreased risk of post-operative sensory loss or neuropathic pain, no need for general anesthesia (local anesthesia) and possible performance on an outpatient basis. By enlarging Physical Medicine and Rehabilitation (PMR) therapeutical armamentarium, percutaneous CN could represent a new compromise between botulinum toxin iterative injections and radical surgery, in terms of invasiveness & complications/long-term benefit ratio on spasticity and function.

The CRYOSTROKE study was designed:

* to compare the efficacy and safety of percutaneous CN versus surgical neurotomy on spasticity, 90 days after intervention, in post-stroke patients presenting with spastic equinovarus foot and,
* to ensure that potential clinical effect/safety remain stable within time, with a 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Patient with spastic equinovarus foot as a result of stroke in chronic phase (>6 months).
* Patient with positive perineural motor block test with or without complete correction of spastic equinus and non-persistence of 40° equinus.
* Patient eligible for surgical neurotomy for varus equinus foot.
* Patient presenting no cognitive impairment or major depression (Mini Mental State Examination>20, Hospital Anxiety and Depression (HAD<11)).
* Absence of active psychosis or history of serious psychotic illness requiring hospitalization
* Patient understanding and accepting the constraints of the study.
* Patient covered by French national health insurance.
* Patient who has given their written consent to the study after having received clear information.

Exclusion Criteria:

* Patient with previous nerve procedures such as chemical neurolysis with alcohol, cryoneurotomy, or any surgery at the same anatomical site.
* Patient with any neurological pathology different from the one responsible for the spasticity.
* Patient with botulinum toxin in lower limb injection during the last 90 days before intervention.
* Patient with anti-spastic treatment (baclofene) up 3 days before block test.
* Patient with total deficit of valgus muscles.
* Patient with equinus foot > 40° (retractions/ankylosis).
* Surgical and anesthetic contra-indications (severe uncontrolled coagulation disorder, active infection).
* Cryoneurotomy contra-indications (cold intolerance, cryoglobulinemia, cryofibrinogenemia, Raynaud's phenomena, venous thromboemolism (< 3 months if superficial, < 6 months if deep), hypothyreosis, cold urticari, local disorders of blood supply, considerable anemia, cachexia, hypothermia, cancer disease, infection, coagulopathy…).).
* Subject requiring closer protection, i.e. minors, pregnant women, nursing mothers, subjects deprived of their freedom by a court or administrative decision, subjects admitted to a health or social welfare establishment, major subjects under legal protection (temporary or permanent guardianship and, subject to subordination), and finally patients in an emergency setting.
* Pregnant woman, nursing mother, woman of childbearing potential not using effective contraception (hormonal/barrier: oral, parenteral, percutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total ovariectomy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2029-04-09 (Estimated); Study Completion 2029-06-09 (Estimated)

PRIMARY OUTCOMES:
Mean absolute change in spasticity assessed by the Modified Ashworth Scale (MAS) ranging from 0 (no spasticity) to 4 (maximum spasticity). | Between baseline and 90-day follow-up
  Mean absolute change in spasticity assessed by the Modified Ashworth Scale (MAS) ranging from 0 (no spasticity) to 4 (maximum spasticity). This MAS will be quantified on a passive ankle dorsal flexion with knee extended (180°) movement.

SECONDARY OUTCOMES:
Mean absolute change in functional disability assessed using the Barthel Index (BI). | Between baseline and 90, 180 and 365-day follow-ups
Mean absolute change in passive ankle dorsal flexion with knee flexed (90°) and extended (180°) movement spasticity assessed by the Modified Ashworth Scale (MAS) | Between baseline and 90, 180 and 365-day follow-ups
Mean absolute change in muscle's response to stretch applied at given velocities assessed by the Tardieu Scale and the Modified Tardieu Scale (MTS) | Between baseline and 90, 180 and 365-day follow-ups
Mean absolute change in maximal ankle range of motion (in degrees) assessed with a goniometer in slow and rapid movement | Between baseline and 90, 180 and 365-day follow-ups
Mean absolute change in the Medical Research Council (MRC) scale of muscle strength of the impaired foot. | Between baseline and 90, 180 and 365-day follow-ups
Mean absolute change in time in seconds to complete the 10-meter walking test | Between baseline and 90, 180 and 365-day follow-ups
Mean absolute change in the distance in meters covered in the 6-min walking test | Between baseline and 90, 180 and 365-day follow-ups
Physical activity intensities: Mean absolute change in the rate of high, moderate, light activities bet | Between baseline and 90, 180 and 365-day follow-ups for a period of 7 days before each visit
Physical activity intensities: mean absolute change in number of steps measured with accelerometer (ActiGraph GT9X) | Physical activity intensities: mean absolute change in number of steps measured with accelerometer (ActiGraph GT9X)
Mean absolute change in pain surface using a digital mapping tool converting pain drawings to cm² | Between baseline and 90, 180 and 365-day follow-ups
Mean absolute change in pain intensity and interference using the Brief Pain Inventory (BPI) questionnaire | Between baseline and 90, 180 and 365-day follow-ups
Mean absolute change in quality of life: EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) questionnaire | Between baseline and 90, 180 and 365-day follow-ups
Mean absolute change in fatigue: Brief Fatigue Inventory (BFI) questionnaire | Between baseline and 90, 180 and 365-day follow-ups
Mean goal attainment assessed with the Goal Attainment Scale (GAS) consisting in 3 main goals provided by the patient before intervention | Between baseline and 90, 180 and 365-day follow-ups
Mean patient satisfaction assessed with Patient Global Impression of Change Patient satisfaction (PGIC) | Between baseline and 90, 180 and 365-day follow-ups
Medico-economic impact measured with Health Care Utilization (HCU) costs | From baseline to 365-day post intervention in terms
Medico-economic impact measured with Employment status | From baseline to 365-day post intervention in terms
Medico-economic impact measured with medication intake | From baseline to 365-day post intervention in terms
Rates of adverse events & serious adverse events | From baseline to 365-day post intervention in terms

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Hôpital Raymond Pointcarré, Garches
  - CHRU Montpellier, Montpellier
  - C.H.U. Poitiers, Poitiers
  - CHU Rennes, Rennes
  - Pôle Saint-Hélier, Rennes
  - CHU Saint-Etienne, Saint-Etienne
  - Hôpital Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: No